CLINICAL TRIAL: NCT00775255
Title: An Open Label, Balanced, Randomised, Two-Treatment, Two-Period, Two-Sequence, Single-Dose, Crossover, Bioavailability Study on Clarithromycin Formulations Comparing Clarithromycin 250 mg/5 mL Powder for Oral Suspension of Ranbaxy Laboratories With Biaxin® Granules 250 mg/5 mL Oral Suspension in Healthy, Adult, Human, Male Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Clarithromycin 250 mg/5 mL Powder for Oral Suspension Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories,
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CPU-M-025/CLARI-250/05
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequiavelnce clarithromycin
MeSH Terms: interventions — Clarithromycin; Powders; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): clarithromycin 250 mg/5 mL powder for oral suspension of Ranbaxy Laboratories
  Interventions: Drug: clarithromycin 250 mg/5 mL powder for oral suspension
- 2 (Active Comparator): Biaxin® granules 250 mg/5 mL oral suspension
  Interventions: Drug: clarithromycin 250 mg/5 mL powder for oral suspension

INTERVENTIONS:
Drug: clarithromycin 250 mg/5 mL powder for oral suspension

SUMMARY:
To compare the single-dose oral bioavailability of clarithromycin 250-mg/5 mL powder for oral suspension of Ranbaxy Laboratories with that of Abbott Laboratories (Biaxin®) following administration of a 250 mg/5 mL dose in healthy, adult, human, male subjects under fasting conditions.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single-dose, crossover, bioavailability study on clarithromycin formulations comparing clarithromycin 250 mg/5 mL powder for oral suspension of Ranbaxy Laboratories with Biaxin® granules 250 mg/5 mL oral suspension (containing clarithromycin 250 mg/5mL) of Abbott Laboratories in healthy, adult, human, male subjects under fasting conditions.

A single oral dose of clarithromycin 250-mg/5 mL was administered during each period of the study under supervision of a trained Medical Officer.

During the course of the study safety parameters assessed were vital signs, twelve-lead ECG, clinical examination, medical history, clinical laboratory safety tests (hematology, biochemical parameters and urine analysis) at base line and hematology and biochemical parameters at 24 hours post dose of the last period of the study. Twelve-lead ECG was recorded at 4 and 8 hours post-dose in each period.

A Validated analytical method was used for the analysis of Clarithromycin in human plasma. Pharmacokinetic and statistical analysis was performed to conclude the bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

1. Be in the age range of 18-45 years.
2. Be neither overweight nor underweight for his/her height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
3. Have voluntarily given written informed consent to participate in this study.
4. Be of normal health as determined by medical history and physical examination of the subjects performed within 14 days prior to the commencement of the study.

Exclusion Criteria:

1. History of allergy to clarithromycin, erythromycin and related macrolides.
2. History of severe diarrhoea within 2 weeks preceding Day 1 of this study.
3. Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
4. Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
5. Presence of values which were significantly different from normal reference ranges (as defined in Appendix 5) and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
6. Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids)
7. Presence of values which were significantly different from normal reference ranges (as defined in Appendix 5) and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
8. Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), glucose (positive) or protein (positive).
9. Clinically abnormal ECG or Chest X-ray.
10. QTc interval beyond normal limits.
11. History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes or glaucoma.
12. History of any psychiatric illness which might have impair the ability to provide written informed consent.
13. Regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
14. History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or have difficulty in abstaining for the duration of each study period.
15. Use of any enzyme modifying drugs within 30 days prior to Day 1 of this study.
16. Participation in any clinical trial within 12 weeks preceding Day 1 of this study.
17. Subjects who, through completion of this study, would have donated and/or lost more than 350 mL of blood in the past 3 months.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2005-09 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Gurgaon, Haryana, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html